CLINICAL TRIAL: NCT03289325
Title: Impact of Perioperative Dexmedetomidine on Long-term Outcomes in Elderly Patients After Cardiac Surgery: 6-year Follow-up of a Randomized Controlled Trial
Brief Title: Dexmedetomidine and Long-term Outcomes in Elderly Patients After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2016-1188
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2023-10

CONDITIONS: Cardiac Surgery; Dexmedetomidine; Long-term Outcome; Mortality; Quality of Life
Keywords: Cardiac surgery; Dexmedetomidine; Long-term outcome; Mortality; Quality of life
MeSH Terms: interventions — Dexmedetomidine; Injections; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEX group (Experimental): The active drug (dexmedetomidine hydrochloride for injection) will be administered during a period from before anesthesia induction until the end of mechanical ventilation after surgery.
  Interventions: Drug: dexmedetomidine hydrochloride for injection
- CTRL group (Placebo Comparator): The placebo drug (normal saline, or 0.9% sodium chloride for injection) will be administered in the same rate and volume for a same duration as that in the DEX group.
  Interventions: Drug: 0.9% sodium chloride for injection

INTERVENTIONS:
Drug: dexmedetomidine hydrochloride for injection — Before anesthesia, dexmedetomidine hydrochloride for injection (200 ug/2 ml) will be diluted with normal saline to 50 ml (final dexmedetomidine concentration 4 ug/ml).
  Before anesthesia induction, a loading dose will be administered by intravenous infusion at a rate of [0.9*kg] ml/h for 10 minutes (i.e., dexmedetomidine 0.6 ug/kg in 10 minutes), followed by continuous infusion at a rate of [0.1*kg] ml/h (i.e., dexmedetomidine at a rate of 0.4 ug/kg/h) until the end of surgery.
  After surgery, the infusion rate will be decreased to [0.025*kg] ml/h (i.e., dexmedetomidine at a rate of 0.1 ug/kg/h) and continued until the end of mechanical ventilation.
  Other Names: Aibeining (trade name)
  Arms: DEX group
Drug: 0.9% sodium chloride for injection — Before anesthesia, 0.9% sodium chloride for injection 50 ml will be prepared.
  Before anesthesia induction, a loading dose will be administered by intravenous infusion at a rate of [0.9*kg] ml/h for 10 minutes, followed by continuous infusion at a rate of [0.1*kg] ml/h until the end of surgery.
  After surgery, the infusion rate will be decreased to [0.025*kg] ml/h and continued until the end of mechanical ventilation.
  Other Names: Normal saline
  Arms: CTRL group

SUMMARY:
A retrospective study showed that intraoperative dexmedetomidine administration was associated with decreased risk of 1-year mortality after cardiac surgery. In a previous randomized controlled trial, 285 elderly patients undergoing cardiac surgery were randomized to receive either perioperative dexmedetomidine or placebo (normal saline) administration. The purpose of this 6-year follow-up study is to investigate whether perioperative dexmedetomidine can improve long-term outcomes in those recruited elderly patients after cardiac surgery.

DETAILED DESCRIPTION:
Dexmedetomidine is a highly selective alpha 2-adrenergic receptor agonist that provides anti-anxiety, sedation, and modest analgesic effects. In a retrospective cohort study of patients undergoing cardiac surgery, perioperative dexmedetomidine administration was associated with decreased risk of 1-year mortality. Theoretically, perioperative dexmedetomidine may exert the following favorable for cardiac surgery patients: (1) reduces perioperative opioid consumption and thereby mitigates opioid-induced immunosuppression, (2) dampens hyper-inflammatory response induced by surgery, and (3) improves postoperative sleep quality. However, prospective studies investigating the long-term effects of perioperative dexmedetomidine in cardiac surgery patients are still lacking.

In a previous randomized controlled trial, 285 patients of 60 years or older who were scheduled to undergo coronary artery bypass graft surgery and/or valve replacement surgery were randomized to receive either perioperative dexmedetomidine administration (0.6 microgram/kg in 10 minutes before anesthesia induction, followed by a continuous infusion at a rate of 0.4 microgram/kg/h until the end of surgery, then a continuous infusion at a rate of 0.1 microgram/kg/h until the end of mechanical ventilation) or placebo (normal saline, administered in the same rate or volume for the same duration as in the dexmedetomidine group). The results showed that perioperative dexmedetomidine reduced the incidence of pulmonary complications and shortened the duration of mechanical ventilation after surgery.

The purpose of this 6-year follow-up study is to investigate the effects of perioperative dexmedetomidine on the long-term outcomes in elderly patients after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 60 years or older;
2. Scheduled to undergo cardiac surgery (coronary artery bypass graft and/or valve replacement surgery);
3. Provide written informed consents.

Exclusion Criteria: Patients who meet any of the following criteria will be excluded.

1. Preoperative history of schizophrenia, epilepsia, Parkinson syndrome, or severe dementia;
2. Inability to communicate in the preoperative period because of severe visual/auditory dysfunction or language barrier;
3. History of brain injury or neurosurgery;
4. Preoperative sick sinus syndrome, severe bradycardia (HR < 50 bpm), second-degree or above atrioventricular block without pacemaker;
5. Severe hepatic dysfunction (Child-Pugh class C);
6. Severe renal dysfunction (requirement of renal replacement therapy);
7. Other conditions that are considered unsuitable for participation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Overall survival after surgery | Up to 6 years after surgery
  Overall survival after surgery

SECONDARY OUTCOMES:
Major adverse cardiovascular events-free survival after surgery | Up to 6 years after surgery
  Major adverse cardiovascular events include cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, and myocardial revascularization.
Hospital-free survival after surgery | Up to 6 years after surgery
  Event indicates any medical condition that lead to hospitalization after surgery.
Cognitive function in 6-year survivors after surgery | At the 6th year after surgery
  Cognitive function is assessed with Telephone Interview for Cognitive Status-Modified (TICS-M; scores range from 0 to 50, with higher score indicating better cognitive function).
Health related quality of life in 6-year survivors after surgery | At the 6th year after surgery
  Health related quality of life is assessed with the short-form 36-item health survey questionnaire (SF-36). The SF-36 scale measures eight aspects of health status, i.e., physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. It also measures changes of subjective healthy status during the last year (reported health transition). The scores of the above 9 items are calculated separately with scores range from 0 to 100, with higher score indicating better quality.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Fuwai Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guenther U, Radtke FM. Delirium in the postanaesthesia period. Curr Opin Anaesthesiol. 2011 Dec;24(6):670-5. doi: 10.1097/ACO.0b013e32834c7b44. PMID 21971396
- [Background] Morandi A, Pandharipande PP, Jackson JC, Bellelli G, Trabucchi M, Ely EW. Understanding terminology of delirium and long-term cognitive impairment in critically ill patients. Best Pract Res Clin Anaesthesiol. 2012 Sep;26(3):267-76. doi: 10.1016/j.bpa.2012.08.001. PMID 23040280
- [Background] Groen JA, Banayan D, Gupta S, Xu S, Bhalerao S. Treatment of delirium following cardiac surgery. J Card Surg. 2012 Sep;27(5):589-93. doi: 10.1111/j.1540-8191.2012.01508.x. PMID 22978835
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Background] Girard TD, Shintani AK, Ely EW. Comment on "Incidence, risk factors and consequences of ICU delirium" by Ouimet et al. Intensive Care Med. 2007 Aug;33(8):1479-80; author reply 1481-2. doi: 10.1007/s00134-007-0698-8. Epub 2007 Jun 5. No abstract available. PMID 17549453
- [Background] Thomason JW, Shintani A, Peterson JF, Pun BT, Jackson JC, Ely EW. Intensive care unit delirium is an independent predictor of longer hospital stay: a prospective analysis of 261 non-ventilated patients. Crit Care. 2005 Aug;9(4):R375-81. doi: 10.1186/cc3729. Epub 2005 Jun 1. PMID 16137350
- [Background] Milbrandt EB, Deppen S, Harrison PL, Shintani AK, Speroff T, Stiles RA, Truman B, Bernard GR, Dittus RS, Ely EW. Costs associated with delirium in mechanically ventilated patients. Crit Care Med. 2004 Apr;32(4):955-62. doi: 10.1097/01.ccm.0000119429.16055.92. PMID 15071384
- [Background] Hopkins RO, Jackson JC. Short- and long-term cognitive outcomes in intensive care unit survivors. Clin Chest Med. 2009 Mar;30(1):143-53, ix. doi: 10.1016/j.ccm.2008.11.001. PMID 19186286
- [Background] Jackson JC, Gordon SM, Hart RP, Hopkins RO, Ely EW. The association between delirium and cognitive decline: a review of the empirical literature. Neuropsychol Rev. 2004 Jun;14(2):87-98. doi: 10.1023/b:nerv.0000028080.39602.17. PMID 15264710
- [Background] Vaurio LE, Sands LP, Wang Y, Mullen EA, Leung JM. Postoperative delirium: the importance of pain and pain management. Anesth Analg. 2006 Apr;102(4):1267-73. doi: 10.1213/01.ane.0000199156.59226.af. PMID 16551935
- [Background] Halaszynski TM. Pain management in the elderly and cognitively impaired patient: the role of regional anesthesia and analgesia. Curr Opin Anaesthesiol. 2009 Oct;22(5):594-9. doi: 10.1097/ACO.0b013e32833020dc. PMID 19623056
- [Background] Rudolph JL, Ramlawi B, Kuchel GA, McElhaney JE, Xie D, Sellke FW, Khabbaz K, Levkoff SE, Marcantonio ER. Chemokines are associated with delirium after cardiac surgery. J Gerontol A Biol Sci Med Sci. 2008 Feb;63(2):184-9. doi: 10.1093/gerona/63.2.184. PMID 18314455
- [Background] de Rooij SE, van Munster BC, Korevaar JC, Levi M. Cytokines and acute phase response in delirium. J Psychosom Res. 2007 May;62(5):521-5. doi: 10.1016/j.jpsychores.2006.11.013. PMID 17467406
- [Background] Roth-Isigkeit A, Borstel TV, Seyfarth M, Schmucker P. Perioperative serum levels of tumour-necrosis-factor alpha (TNF-alpha), IL-1 beta, IL-6, IL-10 and soluble IL-2 receptor in patients undergoing cardiac surgery with cardiopulmonary bypass without and with correction for haemodilution. Clin Exp Immunol. 1999 Nov;118(2):242-6. doi: 10.1046/j.1365-2249.1999.01050.x. PMID 10540185
- [Background] Holmes JH 4th, Connolly NC, Paull DL, Hill ME, Guyton SW, Ziegler SF, Hall RA. Magnitude of the inflammatory response to cardiopulmonary bypass and its relation to adverse clinical outcomes. Inflamm Res. 2002 Dec;51(12):579-86. doi: 10.1007/pl00012432. PMID 12558191
- [Background] Bidwell J. Interventions for preventing delirium in hospitalized non-ICU patients: A Cochrane review summary. Int J Nurs Stud. 2017 May;70:142-143. doi: 10.1016/j.ijnurstu.2016.11.010. Epub 2016 Nov 17. No abstract available. PMID 28160968
- [Background] Liu C, Zhang Y, She S, Xu L, Ruan X. A randomised controlled trial of dexmedetomidine for suspension laryngoscopy. Anaesthesia. 2013 Jan;68(1):60-6. doi: 10.1111/j.1365-2044.2012.07331.x. Epub 2012 Oct 29. PMID 23106186
- [Background] Gozalo-Marcilla M, Hopster K, Gasthuys F, Hatz L, Krajewski AE, Schauvliege S. Effects of a constant-rate infusion of dexmedetomidine on the minimal alveolar concentration of sevoflurane in ponies. Equine Vet J. 2013 Mar;45(2):204-8. doi: 10.1111/j.2042-3306.2012.00613.x. Epub 2012 Aug 1. PMID 22853551
- [Background] Bekker A, Haile M, Kline R, Didehvar S, Babu R, Martiniuk F, Urban M. The effect of intraoperative infusion of dexmedetomidine on the quality of recovery after major spinal surgery. J Neurosurg Anesthesiol. 2013 Jan;25(1):16-24. doi: 10.1097/ANA.0b013e31826318af. PMID 22824921
- [Background] Shim JJ, Leung JM. An update on delirium in the postoperative setting: prevention, diagnosis and management. Best Pract Res Clin Anaesthesiol. 2012 Sep;26(3):327-43. doi: 10.1016/j.bpa.2012.08.003. PMID 23040284
- [Background] Park JK, Cheong SH, Lee KM, Lim SH, Lee JH, Cho K, Kim MH, Kim HT. Does dexmedetomidine reduce postoperative pain after laparoscopic cholecystectomy with multimodal analgesia? Korean J Anesthesiol. 2012 Nov;63(5):436-40. doi: 10.4097/kjae.2012.63.5.436. Epub 2012 Nov 16. PMID 23198038
- [Background] Anger KE. Dexmedetomidine: a review of its use for the management of pain, agitation, and delirium in the intensive care unit. Curr Pharm Des. 2013;19(22):4003-13. doi: 10.2174/1381612811319220009. PMID 23228319
- [Background] Ji F, Li Z, Nguyen H, Young N, Shi P, Fleming N, Liu H. Response to letters regarding article, "perioperative dexmedetomidine improves outcomes of cardiac surgery". Circulation. 2013 Oct 15;128(16):e339-40. doi: 10.1161/CIRCULATIONAHA.113.005450. No abstract available. PMID 24126331
- [Derived] Hong H, Li X, Yang J, Zhang Y, Liu GY, Yan FX, Wang DX. Impact of perioperative dexmedetomidine on long-term outcomes in older patients following cardiac surgery: follow-up of a randomized trial. BMC Anesthesiol. 2025 Mar 17;25(1):130. doi: 10.1186/s12871-025-02963-w. PMID 40097932